CLINICAL TRIAL: NCT01514617
Title: Diffusion -and Perfusion Weighted MRI for Response Prediction of Symptomatic Leiomyomas Following Uterine Artery Embolization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: S53666
Record Dates: First submitted 2011-10-28; First posted 2012-01-23 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Leiomyomas
Keywords: Leiomyoma; Diffusion weighted MRI; Perfusion MRI; Uterine artery embolization; Volumetric Response; Women with symptomatic leiomyomas
MeSH Terms: conditions — Leiomyoma | interventions — gadoterate meglumine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Diffusion -and perfusion weighted MRI including iv contrast agent injection — MRI is a technique based on magnetic fields and does not require the use of ionizing radiation. Although there are no known side effects associated with MRI, a few precautions should be taken because of the 3T magnetic field. This implicates that all metal and magnetized objects must be removed from the patients before entering the MRI room. Patients with a pacemaker, a cardiac defibrillator or other implanted conductors/prostheses are for reason not eligible for the study.
  During the MRI examination, an intravenous contrast agent will be administered. In most cases, patients do not experience any discomfort and the use of this contrast agent is part of the clinical routine.
  Other Names: Dotarem

SUMMARY:
It is known that volumetric response of leiomyomas following uterine artery embolization correlates well with patients clinical outcome. The aim of this study is to assess diffusion -and perfusion weighted MRI for the prediction of volumetric response following uterine artery embolization in patients with symptomatic leiomyomas.

ELIGIBILITY:
Inclusion Criteria:

* women with symptomatic leiomyomas

Exclusion Criteria:

* women with known contra-indications for MRI (cardiac pacemaker, cochlear implants, claustrophobic patients)
* women with contra-indications to gadolinium-based contrast agents (including patients with a known restricted renal function; GFR < 30 mL/min)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diffusion -and perfusion weighted MRI as a predictor for volumetric response of leiomyomas after uterine artery embolization | Participants will be followed for the duration of hospital stay (an expected average of 3 days) and will be systematically followed during their follow-up.
  Patients will be scanned before (baseline) and after (the day of embolization, 3 days and 3 months after embolization). Measurements of signal intensity (SI) will be performed placing ROIs in the central portion of the lesion avoiding areas of artifact. Apparent diffusion coefficients (ADCs) will be calculated at different time points (before and after embolization). Signal intensity measurements on the dynamic contrast enhanced imaging data sets will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Maleux, MD, Prof., Principal Investigator — University Hospital Gasthuisberg, department of Interventional Radiology
Locations (1):
- Radiology Department, Leuven, Belgium